CLINICAL TRIAL: NCT03047304
Title: Magnesium Effect on Embryonal PR Interval
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Ola Gutzeit MD, Principal investigator, Rambam Health Care Campus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0531-15-RMB
Record Dates: First submitted 2017-02-06; First posted 2017-02-08 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Preterm Labor
MeSH Terms: conditions — Obstetric Labor, Premature

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Women in risk for preterm labor (Other): Women in risk for preterm labor treated with magnesium.
  Interventions: Diagnostic Test: Trans abdominal sonography

INTERVENTIONS:
Diagnostic Test: Trans abdominal sonography — Trans abdominal sonography in order to measure fetal PR interval.

SUMMARY:
Magnesium is a known treatment for neuroprotection in preterm labor before 32 week of gestation. High concentration of Magnesium in the blood stream known as cause of conduction abnormalities and ECG changes such us prolonged QT, QRS and PR in about. The goal of our work is to evaluate the PR intervals in embryos after maternal treatment with magnesium during preterm labor.

DETAILED DESCRIPTION:
We will recruit 25 woman with threaten preterm labor, magnesium blood level and PR interval will be evaluated before magnesium loading dose (4gr) and 20 minutes after the loading dose.

PR interval will be evaluated by Mitral-Aorta Doppler.

ELIGIBILITY:
Inclusion Criteria:

* Women at risk for preterm labor before 32 week of gestation

Exclusion Criteria:

* Fetal malformations
* Maternal Lupus
* Fetal conduction abnormalities

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2017-02-14 (Estimated); Primary Completion 2018-02-10 (Estimated); Study Completion 2018-03-10 (Estimated)

PRIMARY OUTCOMES:
Prolonged PR interval | 20 min after magnesium treatment
  PR will be measured by Mitral-aorta doppler

CONTACTS AND LOCATIONS:
Overall Officials: Ola Gutzeit, MD, Principal Investigator — Principal Investigator

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gums JG. Clinical significance of magnesium: a review. Drug Intell Clin Pharm. 1987 Mar;21(3):240-6. doi: 10.1177/106002808702100301. PMID 3552543
- [Background] Agus ZS, Morad M. Modulation of cardiac ion channels by magnesium. Annu Rev Physiol. 1991;53:299-307. doi: 10.1146/annurev.ph.53.030191.001503. No abstract available. PMID 1710436
- [Background] Laurant P, Touyz RM. Physiological and pathophysiological role of magnesium in the cardiovascular system: implications in hypertension. J Hypertens. 2000 Sep;18(9):1177-91. doi: 10.1097/00004872-200018090-00003. PMID 10994748
- [Background] Glickstein JS, Buyon J, Friedman D. Pulsed Doppler echocardiographic assessment of the fetal PR interval. Am J Cardiol. 2000 Jul 15;86(2):236-9. doi: 10.1016/s0002-9149(00)00867-5. No abstract available. PMID 10913494